CLINICAL TRIAL: NCT03967782
Title: Effect of the Exercise-meal Timing on Energy Intake and Appetite in Adolescents With Obesity: the TIMEX 2 Study
Brief Title: Effect of the Exercise-meal Timing on Energy Intake and Appetite in Adolescents With Obesity
Acronym: TIMEX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: AME2P Laboratory, Clermont Auvergne University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2019 BOIRIE; 2019-A00507-50 (Other: 2019-A00507-50)
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-10

CONDITIONS: Pediatric obésity
Keywords: appetite control; obesity; adolescents; exercise timing
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohorte 1 (Experimental): 18 adolescents with obesity are involved and will perform the three conditions.
  Interventions: Behavioral: CON; Behavioral: EX-MEAL; Behavioral: MEAL-EX

INTERVENTIONS:
Behavioral: CON — Control condition without exercise / rest condition. The adolescents will be asked to remain quiet and at rest during the morning and will receive an ad libitum meal at lunch and dinner times. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
  Other Names: control condition without exercise / rest condition
Behavioral: EX-MEAL — Condition with an acute exercise set right before lunch The adolescents will be asked to complete a 30 minutes exercise set at 65% of their capacities (cycling) right before ad ad libitum lunch meal. Lunch will be served ad libitum as well as diner. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
  Other Names: Condition with an acute exercise set right before lunch
Behavioral: MEAL-EX — . condition with an acute exercise set right after lunch. The adolescents will be asked to complete a 30 minutes exercise set at 65% of their capacities (cycling) right after an ad libitul buffet meal. Lunch will be served ad libitum as well as diner. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
  Other Names: Condition with an acute exercise set right after lunch

SUMMARY:
The aim of the present study is to compare the effect of realizing an exercise right before or right after a meal of on energy intake, appetite feelings and food reward in adolescents with obesity.

DETAILED DESCRIPTION:
The present study will compare the nutritional response to the realisation of an acute exercise right before or right after lunch in adolescents with obesity. 18 adolescents with obesity will be asked to randomly complete three experimental sessions: i) one control session (rest); ii) one session with an acute exercise realized right before lunch; iii) one session with an acute exercise realized right after lunch. Their ad libitum energy intake will be assessed during lunch as well as at dinner time. Appetite feelings will be assessed at regular intervals and their food reward in response to the lunch will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI percentile > 97th percentile according to the french curves.
* ages 12-16 years old
* Signed consent form
* being registered in the national social security system
* no contraindication to physical activity

Exclusion Criteria:

* Previous surgical interventions that is considered as non-compatible with the study.
* Diabetes
* weight loss during the last 6 months
* cardiovascular disease or risks

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2019-08-31 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in energy intake measured during an ad libitum buffet meal (in kcal) | day 1 , day 8, day 15
  food intake will be measured ad libitum during a lunch buffet. The adolescents will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be weighted using an electronic food scale by a member of the investigation team and then analysed using Bilnuts software.

SECONDARY OUTCOMES:
Hunger feelings | day 1 , day 8, day 15
  hunger area under the curve will be assessed using visual analogue scale through a the day
Food reward | day 1 , day 8, day 15
  The participants will be asked to complete a validated computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ) (Finlayson, King et al. 2008).

CONTACTS AND LOCATIONS:
Overall Officials: yves Boirie, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moore H, Pereira B, Fillon A, Miguet M, Masurier J, Beaulieu K, Finlayson G, Thivel D. The association between obesity severity and food reward in adolescents with obesity: a one-stage individual participant data meta-analysis. Eur J Nutr. 2024 Jun;63(4):1241-1255. doi: 10.1007/s00394-024-03348-4. Epub 2024 Feb 20. PMID 38376518
- [Derived] Fillon A, Beaulieu K, Miguet M, Bailly M, Finlayson G, Julian V, Masurier J, Mathieu ME, Pereira B, Duclos M, Boirie Y, Thivel D. Does exercising before or after a meal affect energy balance in adolescents with obesity? Nutr Metab Cardiovasc Dis. 2020 Jun 25;30(7):1196-1200. doi: 10.1016/j.numecd.2020.04.015. Epub 2020 Apr 23. PMID 32482455